CLINICAL TRIAL: NCT07109037
Title: Therapeutic Efficacy of Combined Sling Exercise Therapy and Conventional Exercise Therapy in Adult Idiopathic Scoliosis：A Randomized Controlled Trial
Brief Title: Clinical Study on the Improvement of Adult Idiopathic Scoliosis by Sling Exercise Therapy Training Combined With Conventional Exercise Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Medical University (Other)
Responsible Party: Principal Investigator, Wanlin Zou, Clinical Professor, Southwest Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025001
Record Dates: First submitted 2025-07-24; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Scoliosis; Adult
Keywords: Sling exercise training; Exercise therapy; Adult; Idiopathic scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional exercise therapy group (Active Comparator): Conventional exercise therapy includes four exercises: the "little swallow flying" exercise, the hip bridge exercise, back muscle stretching, and relaxation. It is performed once a day, 45 minutes .
  Interventions: Other: Conventional exercise therapy
- Combined Intervention group (Experimental): Suspension training and conventional exercise therapy
  Interventions: Other: Suspension training and conventional exercise therapy

INTERVENTIONS:
Other: Conventional exercise therapy — Conventional exercise therapy includes four exercises: the "little swallow flying" exercise, the hip bridge exercise, back muscle stretching, and relaxation. It is performed once a day, 45 minutes .
  Arms: Conventional exercise therapy group
Other: Suspension training and conventional exercise therapy — Suspension training alternates with conventional exercise therapy. It is conducted every other day, 45 minutes each time, 2-3 times a week for four consecutive weeks. Elastic ropes for suspension training are chosen based on patients' body mass: single - strand for those with body mass ≤ 30 kg and double - strand for those with body mass > 30 kg. Suspension slings are placed on the head, lower back, and pelvis, and non-elastic rope slings on the ankles. Lower the lifting bed so that the vertical distance from the ankles to the bed surface is about 25-30 cm.
  Arms: Combined Intervention group

SUMMARY:
This study aims to compare the effects of suspension exercise therapy combined with conventional exercise therapy and conventional exercise therapy alone on pain, Cobb angle, functional impairment, and quality of life in adult patients with idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* In the anteroposterior and lateral X-ray films of the spine in the standing position, the Cobb angle is ≥10° and <40°
* The age ranges from 18 to 75 years old
* No previous history of surgery
* Not wearing a corrective brace

Exclusion Criteria:

* Having mental illnesses
* Having severe cognitive and communication disorders
* Having severe cardiopulmonary dysfunction or cardiovascular diseases
* Having adult degenerative and secondary scoliosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Cobb angle | The measurements and evaluations were conducted on the first day of treatment and after the completion of the 30 - day treatment respectively.

SECONDARY OUTCOMES:
Oswestry Disability Index | The evaluation was conducted on the first day of treatment and after the completion of the 30-day treatment respectively.
  The Oswestry Disability Index (ODI) scale consists of 10 dimensions, such as walking, sitting, standing, and self-care ability. Each dimension is scored on a scale from 0 to 5 points, yielding a maximum total score of 50 points and a Minimum total score of 0 points. A higher score on the ODI indicates a more severe degree of functional impairment. The results of the ODI can be classified into four grades: a score range of 0%-20% suggests mild impairment; 21%-40% indicates moderate impairment; 41%-60% represents severe impairment; and 61%-100% reflects extremely severe functional impairment.
Pain score (Visual Analogue Scale, VAS) | The evaluation was conducted on the first day of treatment and after the completion of the 30-day treatment respectively.
  The Visual Analogue Scale（VAS） is a 0-10 scale, with 0 signifying no pain and 10 representing the most excruciating pain one can conceive. When administering the VAS, ensure that the graduated side of the scale is not visible to the patient. Then, ask the patient to mark the point on the ruler that reflects their current pain level. After that, the physician will assign a score according to the marked position. Based on the obtained score, pain can be classified as follows: a score of ≤3 indicates mild pain, 4-6 corresponds to moderate pain, and a score of ≥ 7 represents severe pain.
Quality of life assessment (Scoliosis Research Society - 22 questionnaire, SRS - 22) | The evaluation was conducted on the first day of treatment and after the completion of the 30-day treatment respectively.
  The Scoliosis Research Society-22 (SRS-22) questionnaire was employed to assess the QOL of patients. It evaluates quality of life across five dimensions: functional activities, pain, self -image, psychological state, and treatment satisfaction. Each item is scored from 1 to 5, and the total score, with a maximum of 110 and minimum of 0 , reflects a better QOL as it increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Power-sling suspension device (SPS-F11, Nanjing Sbird Biotechnology Co., Ltd.), Neijiang, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
In order to protect the patients' personal privacy from infringement and to make this part of data available for subsequent research.

REFERENCES:
- [Background] Yildirim S, Ozyilmaz S, Elmadag NM, Yabaci A. Effects of Core Stabilization Exercises on Pulmonary Function, Respiratory Muscle Strength, Peripheral Muscle Strength, Functional Capacity, and Perceived Appearance in Children With Adolescent Idiopathic Scoliosis: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Aug 1;101(8):719-725. doi: 10.1097/PHM.0000000000001984. Epub 2022 Feb 2. PMID 35859288
- [Background] Zhou Z, Liu F, Li R, Chen X. The effects of exercise therapy on adolescent idiopathic scoliosis: An overview of systematic reviews and meta-analyses. Complement Ther Med. 2021 May;58:102697. doi: 10.1016/j.ctim.2021.102697. Epub 2021 Feb 23. PMID 33636298